CLINICAL TRIAL: NCT02922231
Title: Post-Marketing Surveillance (Usage Results Study) of RIXUBIS in Adult and Pediatric Patients With Haemophilia B in South Korea
Status: Completed | Type: Observational
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: 251501
Record Dates: First submitted 2016-09-30; First posted 2016-10-04 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — Factor IX

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- All Study Participants: Participants with congenital hemophilia B (FIX level ≤5%)
  Interventions: Biological: RIXUBIS

INTERVENTIONS:
Biological: RIXUBIS — Recombinant Factor IX (rFIX) for intravenous use
  Other Names: Coagulation Factor IX [Recombinant]; rFIX; BAX326; BAX 326

SUMMARY:
Primary: To characterize the safety of RIXUBIS when used under normal clinical care in South Korea.

Secondary: To describe hemostatic effectiveness in subjects receiving RIXUBIS under normal clinical care in South Korea.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with congenital hemophilia B (FIX level ≤5%)
2. Participant or the participant's legally authorized representative has provided signed informed consent.
3. Participant is indicated for treatment according to the RIXUBIS Korean product leaflet.

Exclusion Criteria:

1. Participants with known hypersensitivity or presence of any contraindication to RIXUBIS or its excipients including hamster protein
2. Participants with Disseminated Intravascular Coagulation (DIC)
3. Participants with signs of fibrinolysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hemophilia B in South Korea who have been prescribed RIXUBIS.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (AEs) | Throughout the study period of approximately 2 years and 6 months
  Seriousness and severity of AEs, including any inhibitory antibody development and/or anaphylactic reactions

SECONDARY OUTCOMES:
Physician rated effectiveness of RIXUBIS for prophylactic treatment in participants <12 years old | Up to 6 months from baseline while on treatment
  Rated on a 4-point ordinal scale: Excellent, Good, Moderate, or none
Participant rated effectiveness of RIXUBIS for prophylactic treatment in participants ≥12 years old | Up to 6 months from baseline while on treatment
  Rated on a 4-point ordinal scale: Excellent, Good, Moderate, or none
Physician rated effectiveness of RIXUBIS for on-demand treatment in participants <12 years old | Up to 6 months from baseline while on treatment
  Rated on a 4-point ordinal scale: Excellent, Good, Moderate, or none
Participant rated effectiveness of RIXUBIS for on-demand treatment in participants ≥12 years old | Up to 6 months from baseline while on treatment
  Rated on a 4-point ordinal scale: Excellent, Good, Moderate, or none

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- South Korea (5):
  - Daegu Catholic University Medical Center, Daegu
  - DaeJeon Eulji University Hospital, Daejeon
  - Chung Hospital, Gyeonggi-do
  - Kim Hugh Chul Internal Medicine, Seoul
  - Korea Hemophilia Foundation, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/